CLINICAL TRIAL: NCT01755221
Title: A Prospective Evaluation of the Utility, Optimal Cutoff and Positive Predictive Value of a Pharyngeal Potential of Hydrogen (pH) Probe for Predicting Proton Pump Inhibitor Response in Treatment Naive Laryngopharyngeal Reflux
Brief Title: Positive Predictive Value of the Dx-pH Probe for Predicting PPI Response in LPR
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: Respiratory Technology Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 71707
Record Dates: First submitted 2012-12-18; First posted 2012-12-24 (Estimated); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Laryngopharyngeal Reflux (LPR); Extraesophageal Reflux; Reflux Laryngitis; Posterior Laryngitis
Keywords: Laryngopharyngeal reflux (LPR); Extraesophageal reflux; Reflux laryngitis; Posterior laryngitis; Proton pump inhibitor (PPI) medication; Restech pH probe
MeSH Terms: conditions — Laryngopharyngeal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adult patients with Reflux Symptom Index scores (RSI) greater than or equal to 13 off PPI therapy: 1. Restech pH probe placement at initial clinic visit; subject returns 24 hrs later for probe removal.
  2. Proton pump inhibitor (PPI) therapy; subject starts PPI medication (omeprazole 40mg once daily) and returns for follow-up visit 8-12 weeks later.
  3. Optional second pH probe placement at follow up visit; Subject returns 24 hours later for probe removal; Subject continues PPI medication for 2 more weeks

SUMMARY:
The purpose of this research study is to better understand whether information obtained from a pH probe can help physicians predict whether a patient will respond to the medication that is prescribed for laryngopharyngeal reflux (LPR). The current treatment given to individuals who are diagnosed with LPR is a course of proton pump inhibitor (PPI) medication. Subjects who agree to participate in this study will have a small flexible tube (about the width of a piece of cooked spaghetti) placed in their throat. This tube measures the pH in the throat over a period of 24 hours and helps physicians study the relationship between pH level, LPR symptoms, and the effectiveness of PPI therapy. This study may help physicians find out if certain symptoms or characteristics can help them predict if the PPI medication will be effective for each patient. After probe removal, subjects will receive compensation. They will return to the clinic at their regularly scheduled follow-up visit with the physician, 8 to 12 weeks after starting the PPI medication. At that time, subjects can choose to participate in an optional probe placement.

DETAILED DESCRIPTION:
The purpose of this research study is to better understand whether information obtained from a pH probe can help physicians predict whether a patient will respond to the medication that is prescribed for laryngopharyngeal reflux (LPR). The current treatment given to individuals who are diagnosed with LPR is a course of proton pump inhibitor (PPI) medication. This medication reduces the amount of gastric acid that is produced and generally leads to symptom relief. In order to study whether the pH probe can help physicians predict if the patient will respond to PPI therapy, the physicians will measure the pH level of patients' throats before they start PPI medication. Subjects who agree to participate in this study will have a small flexible tube (about the width of a piece of uncooked spaghetti) placed in their throat. The physician will place the tube through the nose until the tip is in the back of the throat, high enough so that the patient will not feel it when they talk, eat, drink, or swallow. This tube measures the pH in the throat over a period of 24 hours and helps physicians study the relationship between pH level, LPR symptoms, and the effectiveness of PPI therapy. This study may help physicians find out if certain symptoms or characteristics can help them predict if the PPI medication will be effective for each patient. After probe removal, subjects will receive compensation. They will return to the clinic at their regularly scheduled follow-up visit with the physician, 8 to 12 weeks after starting the PPI medication. At that time, subjects can choose to participate in an optional probe placement.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting for evaluation for symptoms classically associated with LPR with a Reflux Symptom Index (RSI) of greater than or equal to 13. The most common symptoms associated with LPR include hoarseness, throat clearing, globus sensation, nocturnal laryngospasm, postnasal drip, chronic cough, and dysphagia.
* Symptom duration of greater than 1 month
* Ages 18-89

Exclusion Criteria:

* Pre-existing PPI therapy for any indication within two weeks of Dx-pH probe placement visit
* Presence of findings of alternative diagnosis explaining symptoms e.g.: laryngeal mass, objective post nasal drainage
* Contraindication to PPI therapy (i.e.: atrophic gastritis, liver problems, severe bloody diarrhea from antibiotics, osteoporosis, broken bone) or unwillingness to initiate PPI therapy
* Pregnancy: There is no contraindication for the Restech pH probe and pregnancy; however, PPI use in pregnant women is contraindicated and thus pregnant women would be ineligible to participate in this study because they would be unable to complete a course of omeprazole.
* Unwillingness or inability to undergo 24 hour pharyngeal pH probe monitoring (for example, oxygen wearing requirement that prevents probe placement or anatomical preclusions like septal perforation).
* Bleeding disorder and/or unable to stop use of anticoagulants such as aspirin, Coumadin (warfarin), and/or Plavix (clopidogrel)

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People receiving care at Northwestern Medicine for laryngeal symptoms
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2012-08; Primary Completion 2014-11 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
RSI Score | 8-12 weeks after initial clinic visit
  Change from baseline in RSI score at 8-12 weeks after initial clinic visit/initiation of treatment will be used to define a response to PPI therapy
Global improvement in self-reported symptoms | 8-12 weeks after initial clinic visit
  Change from baseline in global improvement in self-reported symptoms at 8-12 weeks after initial clinic visit/initiation of treatment will be used to define response to PPI therapy

SECONDARY OUTCOMES:
Differences in pH between PPI responders and non-responders | 8-12 weeks after initial clinic visit
  The Ryan score, total time (as a percent) and number of events below a pH of 4, 5, 6, and 7 will be compared between PPI responders and non-responders.
Effects of PPI therapy on reflux events | 8-12 weeks after initial clinic visit
  All subjects will have the option of a second pH probe placement at the follow up clinic visit 8-12 weeks after the initial clinic visit to assess the effects of PPI therapy on reflux events.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Tan, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Medical Faculty Foundation (NMFF) Sinus and Allergy Center, Chicago, Illinois, United States

REFERENCES:
- [Background] Branski RC, Bhattacharyya N, Shapiro J. The reliability of the assessment of endoscopic laryngeal findings associated with laryngopharyngeal reflux disease. Laryngoscope. 2002 Jun;112(6):1019-24. doi: 10.1097/00005537-200206000-00016. PMID 12160267
- [Background] Belafsky PC, Postma GN, Koufman JA. Validity and reliability of the reflux symptom index (RSI). J Voice. 2002 Jun;16(2):274-7. doi: 10.1016/s0892-1997(02)00097-8. PMID 12150380
- [Background] Belafsky PC, Postma GN, Koufman JA. Laryngopharyngeal reflux symptoms improve before changes in physical findings. Laryngoscope. 2001 Jun;111(6):979-81. doi: 10.1097/00005537-200106000-00009. PMID 11404607
- [Background] Williams RB, Szczesniak MM, Maclean JC, Brake HM, Cole IE, Cook IJ. Predictors of outcome in an open label, therapeutic trial of high-dose omeprazole in laryngitis. Am J Gastroenterol. 2004 May;99(5):777-85. doi: 10.1111/j.1572-0241.2004.04151.x. PMID 15128336
- [Background] Kawamura O, Aslam M, Rittmann T, Hofmann C, Shaker R. Physical and pH properties of gastroesophagopharyngeal refluxate: a 24-hour simultaneous ambulatory impedance and pH monitoring study. Am J Gastroenterol. 2004 Jun;99(6):1000-10. doi: 10.1111/j.1572-0241.2004.30349.x. PMID 15180717
- [Background] Ali T, Roberts DN, Tierney WM. Long-term safety concerns with proton pump inhibitors. Am J Med. 2009 Oct;122(10):896-903. doi: 10.1016/j.amjmed.2009.04.014. PMID 19786155
- [Background] Friedman M, Hamilton C, Samuelson CG, Kelley K, Taylor R, Darling R, Taylor D, Fisher M, Maley A. The value of routine pH monitoring in the diagnosis and treatment of laryngopharyngeal reflux. Otolaryngol Head Neck Surg. 2012 Jun;146(6):952-8. doi: 10.1177/0194599812436952. Epub 2012 Feb 2. PMID 22301104
- [Background] Ayazi S, Lipham JC, Hagen JA, Tang AL, Zehetner J, Leers JM, Oezcelik A, Abate E, Banki F, DeMeester SR, DeMeester TR. A new technique for measurement of pharyngeal pH: normal values and discriminating pH threshold. J Gastrointest Surg. 2009 Aug;13(8):1422-9. doi: 10.1007/s11605-009-0915-6. Epub 2009 May 7. PMID 19421822
- [Background] Becker V, Graf S, Schlag C, Schuster T, Feussner H, Schmid RM, Bajbouj M. First agreement analysis and day-to-day comparison of pharyngeal pH monitoring with pH/impedance monitoring in patients with suspected laryngopharyngeal reflux. J Gastrointest Surg. 2012 Jun;16(6):1096-101. doi: 10.1007/s11605-012-1866-x. Epub 2012 Mar 27. PMID 22450948
- [Result] Yadlapati R, Pandolfino JE, Lidder AK, Shabeeb N, Jaiyeola DM, Adkins C, Agrawal N, Cooper A, Price CP, Ciolino JD, Gawron AJ, Smith SS, Bove M, Tan BK. Oropharyngeal pH Testing Does Not Predict Response to Proton Pump Inhibitor Therapy in Patients with Laryngeal Symptoms. Am J Gastroenterol. 2016 Nov;111(11):1517-1524. doi: 10.1038/ajg.2016.145. Epub 2016 Apr 19. PMID 27091320
- [Result] Yadlapati R, Adkins C, Jaiyeola DM, Lidder AK, Gawron AJ, Tan BK, Shabeeb N, Price CP, Agrawal N, Ellenbogen M, Smith SS, Bove M, Pandolfino JE. Abilities of Oropharyngeal pH Tests and Salivary Pepsin Analysis to Discriminate Between Asymptomatic Volunteers and Subjects With Symptoms of Laryngeal Irritation. Clin Gastroenterol Hepatol. 2016 Apr;14(4):535-542.e2. doi: 10.1016/j.cgh.2015.11.017. Epub 2015 Dec 9. PMID 26689899